CLINICAL TRIAL: NCT07104110
Title: An Open-Label, Multicenter Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of QLH12016 in Combination With Novel Hormonal Agent in Subjects With Advanced Prostate Cancer
Brief Title: Study of QLH12016 in Combination With Novel Hormonal Agent in Subjects With Advanced Prostate Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLH12016-201
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; enzalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLH12016+NHA (Experimental)
  Interventions: Drug: QLH12016; Drug: abiraterone acetate; Drug: enzalutamide

INTERVENTIONS:
Drug: QLH12016 — oral AR PROTAC
Drug: abiraterone acetate — oral CYP17 inhibitor
Drug: enzalutamide — oral androgen receptor inhibitor

SUMMARY:
This study is designed to determine if experimental treatment with QLH12016 in combination with novel hormonal agent (NHA) is safe, tolerable, and has anti-cancer activity in patients with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form.
* Male, aged ≥ 18 years.
* Life expectancy ≥ 3 months.
* Histologically or cytologically confirmed prostate adenocarcinoma.
* Metastatic prostate cancer.
* Organ function meet protocol requirements.
* Recovered from all reversible AEs related to previous anticancer treatments.

Exclusion Criteria:

* Previous treatment with the following drugs:

  1. AR PROTAC class drugs.
  2. Other systemic anticancer therapy within 3 weeks or 5 half-lives prior to the first administration of the study treatment.
  3. Taditional Chinese medicine with anti-tumor indications within 2 weeks prior to the first administration of the study treatment.
  4. Drugs that may cause drug-drug interactions (DDI) with the study treatment.
  5. Drugs known to prolong the QT interval or potentially cause torsades de pointes ventricular tachycardia
* Presence of central nervous system metastases, leptomeningeal metastasis, or spinal cord compression.
* Radiation therapy involving more than 25% of bone marrow within 4 weeks prior to the first administration of the investigational medicinal product; local radiation therapy within 2 weeks prior to the first administration of the investigational medicinal product.
* Treatment with other investigational drugs or major surgery within 4 weeks.
* Inability to swallow, chronic diarrhea, intestinal obstruction, or other factors affecting drug intake and absorption.
* With severe cardiovascular or cerebrovascular diseases or related history.
* Active, uncontrolled infections.
* History of other significant malignancies within 5 years.
* Moderate to severe pulmonary disease significantly affecting lung function.
* According to the investigator's judgment, there are comorbidities that seriously endanger subject safety or affect the subject's ability to complete the study.
* Allergy to any of the investigational medicinal products or their components.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with adverse events/serious adverse events (Phase Ib) | Throughout phase Ib (approximately 1 year)
  Number of patients with adverse events and with serious adverse events including abnormal clinical observations, abnormal ECG parameters, abnormal laboratory assessments and abnormal vital signs that changed from baseline
The number of subjects with dose-limiting toxicity (DLT), as defined in the protocol (Phase Ib) | From first dose of study treatment until the end of Cycle 1.
  A DLT occurs during Cycle 1 (the DLT assessment period) that is assessed as related to study treatment.
Recommended phase II dose (RP2D) (Phase Ib) | Throughout phase Ib (approximately 1 year)
  RP2D will be selected upon safety, PK and efficacy data.
Objective Response Rate (ORR) (Phase II) | From time of Informed Consent to confirmed progressive disease (approximately 1 year)
  Best response until progression, as defined by RECIST 1.1 and PCWG3
Objective Response Rate (ORR) (Phase II) | From time of Informed Consent to confirmed progressive disease (approximately 1 year).
  Proportion of subjects with ≥ 50% PSA decrease